CLINICAL TRIAL: NCT02982291
Title: Focused Spinal Stenosis Rehabilitation Program vs. Generic Williams Flexion Protocol
Brief Title: Focused Spinal Stenosis Rehabilitation Program for Lumbar Spinal Stenosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting patients
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-182
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Spinal Stenosis Lumbar

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard (Active Comparator)
  Interventions: Procedure: Williams flexion protocol
- Individualized (Experimental)
  Interventions: Procedure: Focused spinal stenosis rehabilitation

INTERVENTIONS:
Procedure: Williams flexion protocol — The Williams flexion protocol group will participate in 15 treatment sessions.
  Arms: Standard
Procedure: Focused spinal stenosis rehabilitation — The focused spinal stenosis rehabilitation group will participate in 5 treatment sessions.
  Arms: Individualized

SUMMARY:
Lumbar spinal stenosis with neurogenic claudication is a common condition in the elderly population and is characterized by bilateral buttock, thigh, or calf discomfort and/or pain, as well as by weakness precipitated by walking and prolonged standing. Self-management options include physical therapy, which includes exercise as a core component for improving the flexibility and mobility of the spine and hips. A Williams flexion protocol has historically been used to treat low-back pain following degenerative changes to the posterior elements of the lumbar spine. However, few studies have been done to validate the efficacy of this protocol. A more focused treatment protocol may be more efficacious. Patients in this study will be randomized to receive either the generic physical therapy protocol (15 sessions) or the focused rehabilitation program (5 sessions). The sessions will take place over the course of 6 months. Outcomes will be assessed using validated questionnaires and physical function tests.

ELIGIBILITY:
Inclusion Criteria:

* Lumbar spinal stenosis with neurogenic claudication
* Symptoms present for at least 3 months
* Moderate to severe acquired or congenital LSS based on radiological evaluation
* Lumbar MRI obtained within the past 12 months prior to initial physical therapy visit
* 40 years of age or older
* Body mass index less than or equal to 35
* Can tolerate a 6-min treadmill test
* Willing to comply with home exercises as prescribed

Exclusion Criteria:

* Acute disc herniation
* Grade 3 or greater spondylolisthesis
* Rheumatoid or autoimmune conditions (e.g., ankylosing spondylitis)
* Active spinal compression fractures
* Knee surgery in the previous 6 months (e.g., total knee arthroplasty)
* Previous spinal fusion
* Absence of pedal pulses
* Inflammation/infectious process
* Myelopathy
* Psychiatric disorder preventing informed consent or participation in assigned physical therapy sessions
* Patients with pending litigation or workers compensation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Change in functional ability | Up to 1 year after initial physical therapy visit
  Change in functional ability will be assessed using the Oswestry Disability Index. The minimum clinically important difference of the ODI has been documented in the literature as a 13-point change.

SECONDARY OUTCOMES:
Pain | Up to 1 year after initial physical therapy visit
  Pain will be measured by the Numerical Pain Rating Scale, on a 0-10 scale, where 0=no pain and 10=worst pain.
Quality of life | Up to 1 year after initial physical therapy visit
  Quality of life will be measured using the PROMIS Physical Function 10a Questionnaire.
Tolerance to exercise | Up to 1 year after initial physical therapy visit
  The Timed Treadmill Test, which requires patients to walk on a treadmill at 1.2 miles per hour and a 1% grade and report when they begin experiencing typical exercise-induced symptoms, will be used.
Physical ability | Up to 1 year after initial physical therapy visit
  Physical ability will be assessed upon exams that measure balance, hip abductor strength, range of motion, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Turner, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States